CLINICAL TRIAL: NCT01894789
Title: ComPArison of the Effect of Ticagrelor Versus Clopidogrel on Myocardial Blood Flow (MBF) and Reserve (MBFR) Measured With Positron Emission TomograpHy (PET) in Patients With Coronary Artery Disease (CAD): The PATH Study
Brief Title: Ticagrelor vs Clopidogrel Effect on MFR in CAD Population
Acronym: PATH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Terrence Ruddy, Dr. Terrence Ruddy, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20130105-01H
Record Dates: First submitted 2013-02-27; First posted 2013-07-10 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Coronary Artery Disease
Keywords: myocardial blood flow; myocardial perfusion imaging; myocardial blood flow reserve; positron emission tomography; adenosine; ticagrelor; clopidogrel
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- stable CAD management (Experimental): Experimental: Ticagrelor (BrilintaTM) 90 mg tablet by mouth twice a day
  Interventions: Drug: Ticagrelor; Drug: Clopidogrel
- CAD comparison group (Active Comparator): Active comparator: clopidogrel 75 mg plus placebo tablet by mouth twice a day.
  Interventions: Drug: Ticagrelor; Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Blinded administration of ticagrelor for 10 days
  Other Names: BrilintaTM
Drug: Clopidogrel — Blinded administration of clopidogrel and placebo for 10 days

SUMMARY:
Ticagrelor is one of 3 anti-platelet medications used in patients with acute coronary syndrome (ACS) to prevent further clot formation and further ischemic damage to myocardial tissue. Overall benefits of one drug over the other is neutral in this generally unstable population. In pre-clinical trials, ticagrelor showed secondary effects, involving the release of adenosine to heart muscle where the demand for blood was increased due to a stress condition. Blood flow was increased, potentially preventing potential damage.

This study will compare ticagrelor, currently only approved for use in ACS patients, against clopidogrel by measuring the myocardial blood flow(MBF) during stress to validate this phenomenon. The effect on blood flow will be measurable by using two specific doses of adenosine as the pharmacologic stress and correlating with measurements of blood flow using positron emission tomography (PET) nuclear imaging.

This study hypothesizes that the increase in MBF during intermediate dose adenosine infusion will be greater in ticagrelor treated subjects compared to clopidogrel treated subjects

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Stable coronary artery disease on stable medical treatment.
3. BMI equal to or less than 30 kg/m2
4. No clinically significant abnormalities in baseline laboratory work
5. No clinically significant arrhythmias on baseline 12-lead electrocardiogram
6. Female subjects must be post-menopausal, surgically sterilized or have negative urine beta human chorionic gonadotropin pregnancy test at initial screening and maintain effective contraceptive methods throughout the trial and for 7 days following the end of dosing treatment.

Exclusion Criteria:

1. Any contraindication against the use of clopidogrel, ticagrelor and/or ASA.
2. Oral anticoagulation therapy.
3. History of intracranial bleeding.
4. Recent or active pathological bleeding, such as peptic ulcer.
5. Moderate or severe hepatic impairment.
6. History or risk of bradycardia.
7. Known second- or third-degree AV block without pacemaker
8. Dyspnea (NYHA III/IV), wheezing asthma or COPD.
9. Coronary artery bypass graft (CABG) surgery within 90 days prior to screening or at any time after consent.
10. Percutaneous coronary intervention (PCI) within 90 days prior to screening or at any time following consent.
11. Acute myocardial infarction or acute coronary syndrome within 60 days prior to screening or at any time following consent.
12. Any scheduled surgery during the trial period, including dental.
13. Concomitant therapy with strong cytochrome CYP 3A inhibitor or inducer.
14. Recent use of dipyridamole, dipyridamole-containing medications (e.g. Aggrenox)
15. Known hypersensitivity to the investigational drug or any of its components.
16. Known hypersensitivity to adenosine.
17. Lactose intolerance
18. Breastfeeding or pregnancy.
19. Claustrophobia or inability to lie still in a supine position
20. Unwillingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Differences in rest MBF, stress MBF and MBFR between ticagrelor and clopidogrel treated patients as measured by PET | q 2 weeks blood flow measurements
  Blinded study drug will be administered for 10 days after which the subject will undergo MPI imaging to measure MBF. The crossover to the other study arm will occur and the study procedure repeated.
  Actual study drug effect will not be known until the study has completed and the treatment unblinded.

SECONDARY OUTCOMES:
The effect of ticagrelor on rest MBF, stress MBF and MBFR will be compared in the normal versus abnormal segments on a segmental and patient basis in the ticagrelor treated subjects | q 2 weeks blood flow measurements
  Blinded study drug will be administered for 10 days after which the subject will undergo MPI imaging to measure rest/stress MBF and myocardial blood flow reserve. The crossover to the other study arm will occur and the study procedure repeated.
  Actual study drug effecting flow will not be known until the study has completed and the treatment unblinded.

CONTACTS AND LOCATIONS:
Overall Officials: Terrence Ruddy, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Pelletier-Galarneau M, Hunter CRRN, Ascah KJ, Beanlands RSB, Dwivedi G, deKemp RA, Chow BJW, Ruddy TD. Randomized Trial Comparing the Effects of Ticagrelor Versus Clopidogrel on Myocardial Perfusion in Patients With Coronary Artery Disease. J Am Heart Assoc. 2017 May 2;6(5):e005894. doi: 10.1161/JAHA.117.005894. PMID 28465300